CLINICAL TRIAL: NCT00263653
Title: Study to Evaluate the Safety, Reactogenicity & Immunogenicity of a Booster Dose of GSK Biologicals' Hib-MenC Given With Priorix™, vs Hib-MenC or Priorix™ Only, in Toddlers (13-14 m) Primed With 3 Doses of Hib (as Part of a DTPa -Containing Vaccine) & MenC-CRM197 Conjugate Vaccines.
Brief Title: Safety, Reactogenicity & Immunogenicity Study to Evaluate a Booster Dose of GSK Biologicals' Hib-MenC Given With Priorix™ in Toddlers (13-14 m) Primed With 3 Doses of Hib and MenC-CRM197
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 103954
Record Dates: First submitted 2005-12-08; First posted 2005-12-09 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Haemophilus Influenzae Type b; Neisseria Meningitidis
MeSH Terms: conditions — Haemophilus Infections | interventions — Vaccines

INTERVENTIONS:
Biological: Haemophilus influenzae type b- and meningococcal (vaccine)

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity and immunogenicity of a booster dose of the candidate Hib-MenC conjugate vaccine given concomitantly with measles, mumps and rubella (MMR) vaccine, versus Hib-MenC only and MMR only, when given to healthy subjects aged 13 to 14 months who were primed with 3 doses of Hib (as part of a DTPa -containing vaccine) and MenC-CRM197.

DETAILED DESCRIPTION:
This multicenter study is open with respect to the treatment allocation, but double-blind with respect to the Hib-MenC-TT lots (3 lots). Hib-MenC-TT and Priorix™, when given separately, serve as active controls. Two blood samples are taken: before and one month after vaccination. Additional vaccines are offered at study end in order to complete the vaccine schedule recommended in Spain

ELIGIBILITY:
Inclusion criteria:

* Healthy male or female between, and including, 13 and 14 months of age.
* Previously completed 3-dose primary vaccination with a MenC-CRM197 vaccine, and Hib (given as part of a combined DTPa-containing vaccine) with at least 6 months between the administration of the third doses and the study entry.

Exclusion criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the study vaccine, or planned use during the study period.
* Previous vaccination against OR history of H. influenzae type b (Hib) and/or meningococcal serogroup C disease and/or measles, mumps or rubella OR known exposure to measles, mumps or rubella within 30 days prior to the start of the present study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of any neurologic disorders or seizures.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine including neomycine

Ages: 13 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 297 (Actual)
Dates: Start 2005-03; Primary Completion 2005-03 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Any grade 3 solicited symptoms (d 0 - 3)

SECONDARY OUTCOMES:
Sol (d 0-3, local & general), unsol & MMR specific (d 0-42) symptoms. SAEs (whole study). Subjects with Hib-MenC (pre&42 d post vacc): SBA-MenC titers, anti-PRP, -PSC conc. Subjects with MMR (42 d post vacc): anti-measles, -mumps, -rubella seroconversion

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- Spain (14):
  - GSK Investigational Site, Almería
  - GSK Investigational Site, Antequera/Málaga
  - GSK Investigational Site, Aravaca
  - GSK Investigational Site, Blanes
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Lleida
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Mollet Del Valles/Barcelona
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Sant Adriá de Beyós, Barcelona
  - GSK Investigational Site, Sant Eugenia de Berga, Barcelona
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Vélez-Málaga

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Carmona A, Miranda M, Barrio F, De Vicente A, Mares J, Munoz E, Diez-Delgado J, Alonso A, Gimenez-Sanchez F, Merino J, Garcia-Corbeira P, Maechler G, Boutriau D; Spanish 103954 Study Group. Reactogenicity and immunogenicity of combined Haemophilus influenzae type b-meningococcal serogroup C conjugate vaccine booster dose coadministered with measles, mumps, and rubella vaccine. Pediatr Infect Dis J. 2010 Mar;29(3):269-71. doi: 10.1097/INF.0b013e3181c15977. PMID 19952860
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 103954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 103954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 103954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 103954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 103954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 103954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register